CLINICAL TRIAL: NCT00962962
Title: Exercise Dose-Response Effects in Prediabetes: Responses and Mechanisms
Brief Title: Exercise Dose-Response Effects in Prediabetes
Acronym: STRRIDE-PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: Pro00012628; R01DK081559 (NIH)
Record Dates: First submitted 2009-08-19; First posted 2009-08-20 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2013-09

CONDITIONS: Pre-Diabetes
Keywords: Abnormal fasting glucose
MeSH Terms: conditions — Glucose Intolerance | interventions — Exercise; Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Low-Amount/Moderate Intensity Exercise (Other): Aerobic exercise at 50% peak oxygen use/consumption expending approximately 1,000 calories per week equaling approximately 10 miles per week OR 2.5-3.5 hours per week
  Interventions: Behavioral: Aerobic Exercise
- High-Amount/Moderate-Intensity Exercise (Other): Aerobic exercise at 50% peak oxygen use/consumption expending approximately 1,600 calories per week equaling approximately 16 miles per week OR 4-6 hours per week
  Interventions: Behavioral: Aerobic Exercise
- High-Amount/Vigorous-Intensity Exercise (Other): Aerobic exercise at 75% peak oxygen use/consumption expending approximately 1,600 calories per week equaling approximately 16 miles per week OR 2-3 hours per week
  Interventions: Behavioral: Aerobic Exercise
- Low-Amount/Moderate-Intensity Exercise + Diet (Other): * Exercise - 150 minutes per week (30 minutes / 5 days per week) of aerobic exercise at 50% peak oxygen use/consumption equaling approximately 10 miles per week
  * Diet - The CLI sessions will provide training on needed skills (e.g., calorie counting, portion size estimation) as well as motivation and support in a group counseling setting designed to achieve a weight loss goal of 5 to 7% of baseline body weight.
  Interventions: Behavioral: Exercise and Diet

INTERVENTIONS:
Behavioral: Aerobic Exercise — Aerobic exercise at 50% peak oxygen use/consumption expending approximately 1,000 calories per week equaling approximately 10 miles per week OR 2.5-3.5 hours per week
  Arms: Low-Amount/Moderate Intensity Exercise
Behavioral: Aerobic Exercise — Aerobic exercise at 50% peak oxygen use/consumption expending approximately 1,600 calories per week equaling approximately 16 miles per week OR 4-6 hours per week
  Arms: High-Amount/Moderate-Intensity Exercise
Behavioral: Aerobic Exercise — Aerobic exercise at 75% peak oxygen use/consumption expending approximately 1,600 calories per week equaling approximately 16 miles per week OR 2-3 hours per week
  Arms: High-Amount/Vigorous-Intensity Exercise
Behavioral: Exercise and Diet — * Exercise - 150 minutes per week (30 minutes / 5 days per week) of aerobic exercise at 50% peak oxygen use/consumption equaling approximately 10 miles per week
  * Diet - The Clinical Lifestyle Intervention sessions will provide training on needed skills (e.g., calorie counting, portion size estimation) as well as motivation and support in a group counseling setting designed to achieve a weight loss goal of 5 to 7% of baseline body weight.
  Arms: Low-Amount/Moderate-Intensity Exercise + Diet

SUMMARY:
The purpose of the study is to evaluate the effects of different amounts and intensities of aerobic exercise training programs, with and without weight loss, in people who are at risk for diabetes. An additional purpose of the study is to evaluate the factors in the blood and in exercising muscles that contribute to the improvement in those risk factors. This information will be used to improve exercise training guidelines for improving cardiovascular and metabolic health in people with abnormal fasting glucose, also known as prediabetes.

DETAILED DESCRIPTION:
729 subjects were consented, 288 participants were randomized.

ELIGIBILITY:
Inclusion Criteria:

* Age: 45-75 years
* Moderately Overweight determined by Body Mass Index: 25.0 - 35.4
* Fasting plasma glucose: > 95 - < 126 mg/dL until 2/15/2012 when lower limit was adjusted to > 100 mg/dL

  o Readings from two separate days, both being > 95 (> 100 after 2/15/2012)and one of the two being < 126
* Low density (LDL) cholesterol: < 190 mg/dL
* Triglycerides: < 600 mg/dL
* Resting blood pressure: < 160/90 mmHg
* Inactive: Exercise < one day/week; Peak oxygen consumption: > 18.0 - < 40.0 ml/kg/min until 2/15/2012 when lower limit was adjusted to 12.0 ml/kg/min
* Medications: Stable use of all medications for > three months

Exclusion Criteria:

* Smoker: Tobacco use within the last 12 months
* Dieting or intending to diet
* Use of potential confounding medications, e.g. Niacin containing drugs
* History of diabetes, heart disease or taking medication for those conditions
* History of hypertension (high blood pressure) not controlled with medication
* Pregnant or intending to become pregnant
* Unwillingness to undergo a three month control/run-in period, be randomized to any one of four intervention groups, submit to thigh muscle biopsies and all other study testing or continuously participate in a randomly assigned exercise training or lifestyle intervention program for six months
* Orthopedic limitations, musculoskeletal disease and/or injury
* Allergic to xylocaine (anesthetic or numbing medicine)
* Inability to give blood continuously through a catheter (please notify the study nurse of any difficulty you have experienced in the past when having your blood drawn; the study nurse will determine whether you are excluded for this reason)
* Unwillingness to exercise at least twice per week at the Duke Center for Living Health and Fitness Center during research study staff supervised times

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2009-07; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Fasting Plasma Glucose | 3 month control and 6 months intervention

SECONDARY OUTCOMES:
Measures of Glucose control | 3 month control and 6 month intervention

CONTACTS AND LOCATIONS:
Overall Officials: William E Kraus, MD, Principal Investigator — Duke University
Locations (1):
- Duke Center For Living, Durham, North Carolina, United States

REFERENCES:
- [Derived] Jiang R, Collins KA, Huffman KM, Hauser ER, Hubal MJ, Johnson JL, Williams RB, Siegler IC, Kraus WE. Genome-Wide Genetic Analysis of Dropout in a Controlled Exercise Intervention in Sedentary Adults With Overweight or Obesity and Cardiometabolic Disease. Ann Behav Med. 2024 Apr 11;58(5):363-374. doi: 10.1093/abm/kaae011. PMID 38489667
- [Derived] Bennett WC, Collins KA, Johnson JL, Slentz CA, Willis LH, Bales CW, Huffman KM, Kraus WE. Effects of exercise amount and intensity versus a combined exercise and lifestyle intervention on metabolic syndrome in adults with prediabetes: a STRRIDE-PD randomized trial. Front Physiol. 2023 Jul 14;14:1199763. doi: 10.3389/fphys.2023.1199763. eCollection 2023. PMID 37520827
- [Derived] Sarzynski MA, Ruiz-Ramie JJ, Barber JL, Slentz CA, Apolzan JW, McGarrah RW, Harris MN, Church TS, Borja MS, He Y, Oda MN, Martin CK, Kraus WE, Rohatgi A. Effects of Increasing Exercise Intensity and Dose on Multiple Measures of HDL (High-Density Lipoprotein) Function. Arterioscler Thromb Vasc Biol. 2018 Apr;38(4):943-952. doi: 10.1161/ATVBAHA.117.310307. Epub 2018 Feb 8. PMID 29437573
- [Derived] Bartlett DB, Slentz CA, Connelly MA, Piner LW, Willis LH, Bateman LA, Granville EO, Bales CW, Huffman KM, Kraus WE. Association of the Composite Inflammatory Biomarker GlycA, with Exercise-Induced Changes in Body Habitus in Men and Women with Prediabetes. Oxid Med Cell Longev. 2017;2017:5608287. doi: 10.1155/2017/5608287. Epub 2017 May 31. PMID 28642810
- [Derived] Slentz CA, Bateman LA, Willis LH, Granville EO, Piner LW, Samsa GP, Setji TL, Muehlbauer MJ, Huffman KM, Bales CW, Kraus WE. Effects of exercise training alone vs a combined exercise and nutritional lifestyle intervention on glucose homeostasis in prediabetic individuals: a randomised controlled trial. Diabetologia. 2016 Oct;59(10):2088-98. doi: 10.1007/s00125-016-4051-z. Epub 2016 Jul 15. PMID 27421729